CLINICAL TRIAL: NCT02646397
Title: Comparison of Efficacy and Safety Between Benidipine and Hydrochlorothiazide in Fosinopril Treated Chronic Kidney Disease Patients With Hypertension: a Randomized Controlled Trial
Brief Title: Benidipine and Hydrochlorothiazide in Fosinopril Treated Chronic Kidney Disease Patients With Hypertension
Acronym: BEAHIT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); Zhongda Hospital (Other); Ruijin Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Sichuan Provincial People's Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Changlin Mei, Professor, Director of Division of Nephrology, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZKI-CKD-001
Record Dates: First submitted 2015-12-29; First posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Kidney Disease
Keywords: glomerular filtration rate; hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension | interventions — Fosinopril; benidipine; benidipine hydrochloride; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fosinopril,benidipine combination (Experimental): 254 CKD patients with HTN will take oral tablets of fosinopril (20 mg) plus benidipine (4/8 mg）once daily for 6 months.
  Interventions: Drug: Fosinopril; Drug: Benidipine
- Fosinopril,hydrochlorothiazide combination (Experimental): 254 CKD patients with HTN will take oral tablets of fosinopril (20 mg) plus hydrochlorothiazide (12.5/25 mg）once daily for 6 months.
  Interventions: Drug: Fosinopril; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Fosinopril — Fosinopril is an angiotensin-converting enzyme inhibitor.
  Other Names: Fosinopril Sodium; Squibb Brand of Fosinopril Sodium; Fosinil
Drug: Benidipine — Benidipine is a dihydropyridine-derived calcium channel blocker.
  Other Names: benidipine hydrochloride
  Arms: Fosinopril,benidipine combination
Drug: Hydrochlorothiazide — Hydrochlorothiazide is a diuretic medication.
  Other Names: HCTZ; Dichlothiazide; HydroDIURIL
  Arms: Fosinopril,hydrochlorothiazide combination

SUMMARY:
The purpose of this study is to compare the effect of fosinopril plus benidipine vs. fosinopril plus hydrochlorothiazide on the renal function during the 6-month treatment in CKD patients with HTN.

DETAILED DESCRIPTION:
Patients with chronic kidney dysfunction or injury which affected the health over three months were diagnosed with chronic kidney disease (CKD).China has a high prevalence of CKD.The prevalence, awareness, and treatment of hypertension (HTN) in non-dialysis CKD patients were 67.3%,85.8%, and 81.0%, respectively. The renin-angiotensin system inhibitors (RASI) including angiotensin-converting enzyme inhibitor (ACEI) and angiotensin II type 1 receptor blocker (ARB) have been deeply confirmed to have apparent reno-protective effect in patients with CKD.Co-administration of diuretics and calcium channel blockers (CCBs) with ACEIs or ARBs are the most common combinations. Hydrochlorothiazide plus RASIs are another widely used combination according to the synergetic function of antihypertensive action and offset mutual adverse effects. Until now, no large scale studies have compared the effect of initial treatment with two different combinations of antihypertensive drugs in CKD patients on the progression of kidney disease in China. Studies in the subsets of CKD (diabetes and non-diabetes, micro-albuminuria and macro-albuminuria) are urgently needed.We aimed to conduct a large scale study to compare L/T-type CCB and diuretic on the basis of ACEI in CKD with HTN on renal progression of CKD in China.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with non-dialysis CKD at the enrollment and randomization eGFR≥ 30 ml/min per 1.73 m2 at the enrollment and randomization SBP> 130 mmHg and/or DBP > 80 mmHg at the enrollment and randomization. Patients could not receive more than two antihypertensive medications prior to our enrollment, and should discontinue the prior antihypertensive medications after the enrollment according to the investigators' advice.
2. 24 h proteinuria < 1.5g at the enrollment
3. Patients who signed the informed consent form
4. Baseline serum Cr < 3 mg/dL at the enrollment and randomization

Exclusion Criteria:

1. Hypertensive crisis (SBP > 180 mmHg and/or DBP>110 mmHg)
2. Refractory hypertension (taking > 2 antihypertensive drugs more than a month, SBP still > 160mm Hg or DBP > 100mmHg)
3. Baseline serum Cr > 3 mg/dl, or kidney transplantation
4. Patients diagnosed as severe cardiac arrhythmia (severe extra beats, supraventricular tachycardias, ventricular arrhythmias, or bradyarrhythmias), heart failure, NYHA >Ⅲ, angina, stroke, left ventricular hypertrophy or myocardial infarction within 12 months prior to first visit.
5. Patients diagnosed as cancer or severe sepsis
6. Hematological system disorders: myelodysplastic syndrome, granulocytopenia, hypereosinophilic syndrome, polycythemia, thrombocytopenia, and et al.
7. Restrictive pericarditis
8. Systemic Lupus Erythematous
9. Severe diabetes complications such as diabetic ketoacidosis, hyperosmolar coma, retinopathy, amputation, and et al.
10. Patients diagnosed as hyperkalemia(>5.5mmol/L) within 6 months or at the enrollment
11. Renal artery stenosis or vascular embolism disease
12. Patient is currently pregnant or lactational
13. AST/ALT > three times of the upper limit of standard value at the baseline
14. Any severe allergy of CCB, diuretic or ACE inhibitor
15. History of severe side effects of CCB, diuretic or ACE inhibitor; long-term use of non-steroidal anti-inflammatory drugs
16. Use of other investigational drugs within 30 days or 5 half-lives of last visit, whichever is longer.
17. Other unsuitable patients judged by the investigators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changes in estimated glomerular filtration rate | Changes in eGFR at month 6

SECONDARY OUTCOMES:
Abnormal renal events | From baseline to month 6
  Number of participants with 30% reduction of eGFR, doubling of serum creatinine concentration,end-stage renal disease (eGFR< 15 mL/min/1.73m²) or chronic dialysis.
Changes in 24 hour proteinuria | From baseline to month 6
Changes in mean SBP | From baseline to month 6
Abnornal cardiovascular events | At month 6
  Number of participants with cardiovascular morbidity (nonfatal stroke, non-fatal myocardial infarction, resuscitated sudden cardiac death, unstable angina; and coronary revascularization procedures) and cardiovascular mortality (death due to sudden cardiac death, fatal stroke, fatal myocardial infarction, congestive heart failure or other cardiovascular causes).
Adverse Events | From baseline to month 6
  Number of participants with abnormal laboratory values and/or adverse events that are related to Treatment
Changes in urinary albumin excretion | From baseline to month 6
Changes in mean DBP | From baseline to month 6

CONTACTS AND LOCATIONS:
Overall Officials: Changlin Mei, Study Chair — Division of Nephrology, Shanghai ChangZheng Hospital
Locations (1):
- Department of Nephrology, Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xue C, Zhou C, Yang B, Lv J, Dai B, Yu S, Wang Y, Zhao G, Mei C. Comparison of efficacy and safety between benidipine and hydrochlorothiazide in fosinopril-treated hypertensive patients with chronic kidney disease: protocol for a randomised controlled trial. BMJ Open. 2017 Feb 24;7(2):e013672. doi: 10.1136/bmjopen-2016-013672. PMID 28237959